CLINICAL TRIAL: NCT04253054
Title: Chinese Multi-provincial Cohort Study-Beijing Project
Acronym: CMCS-Beijing
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: CMCS-Beijing 2020
Record Dates: First submitted 2020-01-22; First posted 2020-02-05 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Aging Problems; Smell Disorder; Sleep
MeSH Terms: conditions — Cardiovascular Diseases; Olfaction Disorders | interventions — Heart Disease Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, blood cell and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cardiovascular risk factors — Different level of cardiovascular risk factors, such as aging, hypertension, diabetes, dyslipidemia, smoke, alcohol drink, obesity and et al, associated with genetics, environments and lifestyles
Other: Aging related health problems — Aging related health problems

SUMMARY:
The Chinese Multi-provincial Cohort Study (CMCS)-Beijing project is a sub-study in CMCS participants from Beijing, which intended to investigate the progression and determinants of atherosclerosis and aging related health problems through repeat examinations. Exam 0 to Exam 3 have been conducted during 1992 to 2012. Exam 4 is scheduled in 2020.

ELIGIBILITY:
Inclusion Criteria:

* Participants from CMCS-Beijing
* sign the informed consent

Exclusion Criteria:

* participanting in clinical trials

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants were recruited from the Chinese Multi-provincial Cohort Study-Beijing Project
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
All fatal and nonfatal acute coronary and stroke events | From date of enrollment until the date of first documented event or date of cardiovascular death, whichever came first, assessed at least 5 years
  Acute coronary heart disease events included acute myocardial infarction, sudden death, and other coronary deaths. Acute stroke events included subarachnoid hemorrhage, intracerebral hemorrhage, or cerebral infarction.

SECONDARY OUTCOMES:
New-onset of coronary events | From date of enrollment until the date of first documented event or date of CHD death, whichever came first, assessed at least 5 years
  Acute coronary heart disease events included acute myocardial infarction, sudden death, and other coronary deaths.
New-onset of stroke | From date of enrollment until the date of first documented event or date of stroke death, whichever came first, assessed at least 5 years
  Acute stroke events included subarachnoid hemorrhage, intracerebral hemorrhage, or cerebral infarction.
Total death | From date of enrollment until date of death from all cause, assessed at least 5 years
  All cause death
Cognitive dysfunction | From date of enrollment until date of first documented event, assessed at least 5 years
  Cognitive dysfunction
Olfactory Disorders | From date of enrollment until date of first documented event, assessed at least 5 years
  Olfactory Disorders
Valvular disease | From date of enrollment until the date of first documented event or date of valvular disease death, whichever came first, assessed at least 5 years
  Valvular disease

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, MD, PhD, Principal Investigator — Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart, Lung and Blood Vessel Diseases
Locations (3):
- China (3):
  - Beijing Sijiqing Hospital, Beijing, Beijing
  - Peking University Hospital, Beijing, Beijing
  - Peking University Shougang Hospital, Beijing